CLINICAL TRIAL: NCT06458283
Title: Effıcıency Of Hybrıd Based Sımulatıon Method In Breastfeedıng Educatıon Of Mıdwıfery Students
Brief Title: Effıcıency Of Hybrıd Based Sımulatıon Method In Breastfeedıng Educatıon
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Ebru Çalışkan, PhD Midwifery, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BAP2023/18
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breastfeeding; Training Group, Sensitivity; High Fidelity Simulation Training; Medical Simulation; Standardized Patient
Keywords: simulation based breastfeeding training; breast feeding; midwifery; education; Simulation; Standardized Patient; High Fidelity Simulation Training
MeSH Terms: conditions — Breast Feeding; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Investigation of the effectiveness of scenario-based standardized patient simulation training and breastfeeding management of midwifery students
  Interventions: Other: hiybrid simulation
- Control Group (Experimental): Standard training of midwifery students with low fidelty breast model
  Interventions: Other: control grup

INTERVENTIONS:
Other: hiybrid simulation — The intervention group students were given practical training on breast milk and breastfeeding management in the professional skills laboratory, accompanied by a high-reality simulator accompanied by a scenario, and the control group students were given practical training on breast milk and breastfeeding management in the professional skills laboratory, accompanied by an adult standard patient care model.
  Arms: Experimental Group
Other: control grup — low fidelity simulator
  Arms: Control Group

SUMMARY:
It was planned to determine the effect of hybrid simulation-based breastfeeding training on the practical skills, satisfaction, self-confidence and self-efficacy of the students of the Department of Midwifery, Hamidiye Faculty of Health Sciences, University of Health Sciences

DETAILED DESCRIPTION:
This study was planned to determine the effect of hybrid simulation-based breastfeeding education on the practical skills, satisfaction, self-confidence and self-efficacy of the students of the Department of Midwifery, Hamidiye Faculty of Health Sciences, University of Health Sciences. The research, planned in a randomized controlled experimental design, will be conducted with Istanbul Health Sciences University Hamidiye Health Sciences Faculty midwifery 2nd year students (N: 84). Students participating in the study will be divided into intervention (n: 42) and control (n: 42) groups according to the computer-assisted simple random sampling technique. Both groups will be given 4 hours of theoretical information about breast milk and breastfeeding education before the application. 42 students assigned to the intervention group will receive training with a high-reality simulator fitted to a standard patient, accompanied by a scenario, and 42 students assigned to the control group will receive practice training with an adult standard patient care model. Introductory Information Form, Simulation-Based Learning Evaluation Scale, Student Satisfaction and Self-Confidence in Learning Scale, Self-Efficacy-Sufficiency Scale, Breastfeeding Management Skill Evaluation Form will be applied to the students participating in the research.

As a result of the findings, discussion and conclusions of the study will be written.

It is important to increase the competency level of midwifery students in breastfeeding management in a simulation environment that creates virtual reality, before the care applied on real patients in a clinical environment. It is recommended to integrate high-reality simulators and standard patient methods into the curriculum in the education of midwifery students . This study aims to increase the application skills, satisfaction, self-confidence and self-efficacy levels of midwifery department students with hybrid simulation-based Breastfeeding education, in which two or more simulation types (standard patient and Lactation Simulator) are combined to produce a more realistic simulation experience.

ELIGIBILITY:
Inclusion Criteria:

Having a statement of consent Being a second year midwifery student

Exclusion Criteria:

Wishing to withdraw from the research at any time. Not participating in all simulation applications Incompletely filling out data collection forms

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-11-10 (Estimated)

PRIMARY OUTCOMES:
Self-EffectivenessEfficacy Scale | immediately before simulation
  TThe Self-Efficacy Scale is structured as a 5-point Likert scale consisting of 23 items, with a possible score range of 23 to 115. For each item in the scale, respondents are asked to mark one of the following options: 1) Does not describe me at all, 2) Describes me a little, 3) Neutral, 4) Describes me well, and 5) Describes me very well. Items 2, 4, 5, 6, 7, 10, 11, 12, 14, 16, 17, 18, 20, and 22 are scored in reverse. A higher score indicates a higher perception of overall self-efficacy.
Self-EffectivenessEfficacy Scale | immediately after the simulation application
  The Self-Efficacy Scale is structured as a 5-point Likert scale consisting of 23 items, with a possible score range of 23 to 115. For each item in the scale, respondents are asked to mark one of the following options: 1) Does not describe me at all, 2) Describes me a little, 3) Neutral, 4) Describes me well, and 5) Describes me very well. Items 2, 4, 5, 6, 7, 10, 11, 12, 14, 16, 17, 18, 20, and 22 are scored in reverse. A higher score indicates a higher perception of overall self-efficacy.
Self-EffectivenessEfficacy Scale | 4 weeks after the first simulation application
  The Self-Efficacy Scale is structured as a 5-point Likert scale consisting of 23 items, with a possible score range of 23 to 115. For each item in the scale, respondents are asked to mark one of the following options: 1) Does not describe me at all, 2) Describes me a little, 3) Neutral, 4) Describes me well, and 5) Describes me very well. Items 2, 4, 5, 6, 7, 10, 11, 12, 14, 16, 17, 18, 20, and 22 are scored in reverse. A higher score indicates a higher perception of overall self-efficacy.
Introductory Information Form | immediately before simulation
  In this form, which was created by the researchers based on the literature, the participants' age, the high school they graduated from, the education level of their parents, their willingness to choose the profession, their feeling of belonging to the profession, etc. questions are included. The Introductory Information Form is in a multiple-choice format consisting of 25 questions by scanning the literature by the researchers.
Student Satisfaction and Self-Confidence Scale in Learning | immediately after the simulation application
  The scale is a 13-item measurement tool designed to measure student satisfaction with simulation and self-confidence during practices. It is a 5-point Likert type and is scored as strongly disagree 1, disagree 2, undecided 3, agree 4, strongly agree 5.According to the Turkish adaptation of the scale, the total number of items is 12. This scale measures student satisfaction and self-confidence regarding learning in a simulation environment. The scale consists of two subheadings: "Satisfaction with Current Learning" and "Self-Confidence in Learning." The subheading "Satisfaction with Current Learning" includes 5 items, and the subheading "Self-Confidence in Learning" includes 7 items, with no negatively coded items.
Simulation-Based Learning Assessment Scale | immediately after the simulation application
  The scale has 5 sub-dimensions (nursing process, patient safety, professional information, communication and reflected behavior) and consists of 37 items.All statements on the scale are positive, and there are no negatively coded items. The scale evaluates the essential competencies that a nurse should possess, including the nursing process, patient safety, professional knowledge, communication, and reflective behavior concepts. An increase in the score obtained from the sub-dimensions of the scale indica

SECONDARY OUTCOMES:
BREASTFEEDING MANAGEMENT INFORMATION ATTITUDES AND SKILLS EVALUATION FORM | immediately before simulation
  Form of 40 items: 1 Inadequate (0 points 2. Partially Satisfactory/Needs improvement (1 point): 3. Satisfactory (2 points)
BREASTFEEDING MANAGEMENT INFORMATION ATTITUDES AND SKILLS EVALUATION FORM | 4 weeks after the first simulation application
  Form of 40 items: 1 Inadequate (0 points 2. Partially Satisfactory/Needs improvement (1 point): 3. Satisfactory (2 points)

CONTACTS AND LOCATIONS:
Overall Officials: yasemin aydın kartal, Assoc. Prof, Study Director — SAĞLIK BİLİMLERİ ÜNİVERSİTESİ; Ebru ÇALIŞKAN, PhD.Stu., Principal Investigator — SAĞLIK BİLİMLERİ ÜNİVERSİTESİ
Locations (1):
- Sağlık Bilimleri Üniversitesi Hamidiye, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No